CLINICAL TRIAL: NCT06485414
Title: Investigating the Association Between Central Sensitization and Breathing Pattern Disorders : A STROBE-compliant Cross-sectional Study
Brief Title: Investigating the Association Between Central Sensitization and Breathing Pattern Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyunjoong Kim, Principal investigator, Sahmyook University
Other Study IDs: 1014223-202405-HR-01
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Central Sensitisation
Keywords: central sensitization; breathing pattern disorders; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- central sensitization: Individuals who scored above 40 on the Central Sensitization Inventory for Koreans (CSI-K) assessment.

SUMMARY:
Breathing pattern disorders can cause mechanical, physiological, and psychological issues in the body, contributing to the initiation and chronicity of pain. Therefore, considering breathing patterns is significant in managing chronic pain, yet direct research on central sensitization and breathing pattern disorders remains scant. This study aims to analyze the correlation between central sensitization and breathing pattern disorders in adults by assessing both respiration and pain.

DETAILED DESCRIPTION:
Breathing pattern disorders impact consciousness and the body according to respiratory patterns, leading to physiological, mechanical, and psychological disturbances. Unlike normal breathing patterns facilitated by appropriate diaphragmatic activity, incorrect patterns often exhibit reduced diaphragmatic engagement. Chest breathing patterns are prevalent among chronic pain patients, characterized by limited upper chest segment movement due to prolonged improper respiration without specific pathological symptoms. Fluoroscopy studies reveal flattened and tense diaphragms with diminished relative mobility, implicating accessory and inspiratory muscles more heavily in ventilation. Biologically unsustainable functional breathing patterns correlate with chronic musculoskeletal issues and pain. Prior research establishes associations between inappropriate breathing patterns and chronic lower back pain and scapular dysfunctions. Consequently, managing chronic pain clinically necessitates functional recovery and pain relief, crucial for sustaining daily life. Therefore, researching central adaptations and respiration in chronic pain management is imperative, yet remains insufficiently explored.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above.
* Individuals scoring 40 or above on the Central Sensitization Inventory for Koreans (CSI-K).
* Individuals who consent to the use and publication of their personal information and wish to participate in assessment measurements.

Exclusion Criteria:

* Individuals with pulmonary, cardiac, or respiratory diseases.
* Individuals with severe hypertension, defined as systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg.
* Individuals with cognitive impairments.
* Individuals who express a desire to withdraw from the study during its duration.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants were voluntarily recruited from church members who complained of symptoms of central sensitization and were registered according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-03 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory function | During the assessment period
  This study utilized the Self Evaluation of Breathing Questionnaire (SEBQ) to assess respiratory function. The SEBQ is a self-administered questionnaire designed to measure symptoms and severity associated with respiratory dysfunction. It consists of 25 items, each rated on a 4-point scale (0 = not at all, to 3 = very much so), with a total possible score ranging from 0 to 75. While there is no definitive cutoff score for the SEBQ, experts consider a total score above 25 to indicate a problem with respiratory function. The SEBQ has a test-retest reliability (ICC) of 0.89 and internal consistency (Cronbach's α) of 0.93.

CONTACTS AND LOCATIONS:
Overall Officials: Hyunjoong Kim, PhD, Principal Investigator — Gwangju Health University
Locations (1):
- Honam University, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Undecided